CLINICAL TRIAL: NCT06876675
Title: Multicenter Cohort Study of LORLATINIB-related HYPERLIPIDEMIA in ALK+ Advanced Non-Small Cell Lung Cancer Patients
Brief Title: LORLATINIB-related HYPERLIPIDEMIA in ALK+ Non-Small Cell Lung Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Liang, Chief Physician, Peking University Third Hospital
Other Study IDs: (2024)696-02
Record Dates: First submitted 2024-11-25; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer; Hyperlipidemia
Keywords: NSCLC; Hyperlipidemia; Lorlatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hyperlipidemias | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Lorlatinib — To study hyperlipidemia frequency, levels, impact on cardiovascular events after use of Lorlatinib in NSCLC patients.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of Lorlatinib related hyperlipidemia in NSCLC patients who take Lorlatinib for at least 21 days. The main question it aims to answer is:

* Whether blood lipids have been lowered down to an anticipated level within recommended range after the initial revealed Lorlatinib related hyperlipidemia?
* Will it be harmful to the cardiovascular system when blood lipids were not lowered down to normal levels in these cancer patients treated with Lorlatinib, i.e. major adverse cardiac events (MACE), or instead, carotid artery intima-media thickness.

Participants already taking Lorlatinib as part of their regular medical care for NSCLC will answer online survey questions.

ELIGIBILITY:
Inclusion Criteria:

* Advanced ALK+ NSCLC diagnosed by patholgy and/or cytology
* ECOG 0-2
* Age 18-80 years
* Taken Lorlatinib for at least 20 days
* Signed informed consent.

Exclusion Criteria:

* Treatment with other anti-cancer drugs during Lorlatinib treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC patients with ALK fusion positive who were treated with Lorlatinib as first- or later- line therapy will be enrolled from 10 tertiary hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Alteration from baseline to 2 years after first dose of Lorlatinib: maximum carotid intima-media thickness and coronary CT calcification score. | From first dose of Lorlatinib to 2 years thereafter.
  Maximum carotid intima-media thickness: the higher the worse. It is a value directly determined under carotid ultrasound.
  CT: Computed Tomography Coronary CT calcification score: the higher the worse. It is a value directly determined by coronary calcium scan.

SECONDARY OUTCOMES:
Numbers and Time of Major adverse cardiovascular events in patients with Lorlatinib-related hyperlipidemia. | From first dose of Lorlatinib to at maximum of 10 years thereafter.
Comparison of predictive effect on MACE between change in maximum carotid intima-media thickness and coronary artery calcium score. | From first dose of Lorlatinib to at maximum of 10 years thereafter.

OTHER OUTCOMES:
Blood lipid reduction among different lipid-lowering drugs in treating Lorlatinib-related hyperlipidemia. | From first dose of Lorlatinib to 2 years thereafter.
Impact of lipid-lowering drugs on Lorlatinib efficacy. | From first dose of Lorlatinib to 2 years thereafter.
  The Lorlatinib efficacy is clinically measured as per RECIST1.1. Normally patients receiving Lorlatinib will undergo clinical routine CT scans every 1-2 months. Since this study is an observational study, we do not request the time interval for each round of CT scans-just as good as clinical routine.
  In this study, the Lorlatinib efficacy mainly refers to objective response rate(ORR), progression-free survival(PFS) and overall survival(OS). We aim to compare whether different lipid-lowering drugs may have different Lorlatinib efficacy in this prospective cohort.
Correlation between the duration of lorlatinib-related hyperlipidemia and maximum of carotid intima-media thickness. | From first dose of Lorlatinib to 2 years thereafter.
Objective response rate (ORR) | From first dose of Lorlatinib to 2 years thereafter.
  The Lorlatinib efficacy is clinically measured as per RECIST1.1. Normally patients receiving Lorlatinib will undergo clinical routine CT scans every 1-2 months. Since this study is an observational study, we do not request the time interval for each round of CT scans-just as good as clinical routine.
Progression-free Survival (PFS) | From first dose of Lorlatinib to at maximum of 10 years thereafter.
  The Lorlatinib efficacy is clinically measured as per RECIST1.1. PFS is defined as the time from the first dose of Lorlatinib to disease progression.
  Normally patients receiving Lorlatinib will undergo clinical routine CT scans every 1-2 months. Since this study is an observational study, we do not request the time interval for each round of CT scans-just as good as clinical routine.
Overall Survival (OS) | From first dose of Lorlatinib to at maximum of 10 years thereafter.
  The Lorlatinib efficacy is clinically measured as per RECIST1.1. OS is defined as the time from the first dose of Lorlatinib to the date of death.
  Normally patients receiving Lorlatinib will undergo clinical routine CT scans every 1-2 months. Since this study is an observational study, we do not request the time interval for each round of CT scans-just as good as clinical routine.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
IPD will only be acquired by contacting investigator